CLINICAL TRIAL: NCT05291910
Title: A Study to Assess the Efficacy and Safety of Inetetamab Combined With Anti-PD-1 Monoclonal Antibody and Albumin-Bound Paclitaxel for HER2+ Metastatic Breast Cancer
Brief Title: Inetetamab Combined With Anti-PD-1 Monoclonal Antibody and Albumin-Bound Paclitaxel for HER2+ Metastatic Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Binghe Xu, Director of Breast Cancer Section, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPT-2021-002
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — toripalimab; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inetetamab+ Toripalimab+ Albumin-Bound Paclitaxel (Experimental): Drug: Inetetamab Initial dose of 8 mg/kg over 90 minutes IV infusion, then 6 mg/kg over 30 to 90 minutes IV infusion every three weeks Drug: Toripalimab 240mg intravenously every 3 weeks Drug: Albumin-Bound Paclitaxel 130mg/m2, IV , D1, D8, q3w
  Interventions: Drug: Inetetamab; Drug: Toripalimab; Drug: Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: Inetetamab — Initial dose of 8 mg/kg over 90 minutes IV infusion, then 6 mg/kg over 30 to 90 minutes IV infusion every three weeks
Drug: Toripalimab — 240mg intravenously every 3 weeks
Drug: Albumin-Bound Paclitaxel — 130mg/m2, IV , D1, D8, q3w

SUMMARY:
This is a multi-center, prospective, interventional, single-arm clinical trial. In the study, patients with her2-positive recurrent or metastatic breast cancer who were initially treated were included. The purpose of this study is to evaluate the efficacy and safety of Inetetamab combined with anti-PD-1 monoclonal antibody and albumin-bound paclitaxel for HER2+ Metastatic Breast Cancer.

DETAILED DESCRIPTION:
This is a multi-center, prospective, interventional, single-arm clinical trial. In the study, patients with her2-positive recurrent or metastatic breast cancer who were initially treated were included. The purpose of this study is to evaluate the efficacy and safety of Inetetamab combined with anti-PD-1 monoclonal antibody and albumin-bound paclitaxel for HER2+ Metastatic Breast Cancer.To explore a new concept of anti-HER2 monoclonal antibody combined with immunotherapy in the treatment of recurrent or metastatic breast cancer. The primary end point is progression free survival (PFS). The secondary end points are objective response rate (ORR), Clinical Benefit Rate (CBR) and safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged > 18 years.
2. Pathological diagnosis of HER-2 was positive (definition: immunohistochemical results were + + + or ICH++ with fluorescence in situ hybridization results were positive).
3. Participants must have histologically or cytologically confirmed invasive breast cancer with locally recurrent or radiological evidence of metastatic disease.
4. Patients with locally recurrent inoperable or metastatic HER2-positive breast cancer:

   1. patients with metastatic breast cancer at the time of initial diagnosis, meaning there was no previous history of breast cancer in the past; or
   2. patients with Locally recurrent or metastatic breast cancer, neoadjuvant/adjuvant anti-HER2 therapy has been completed for ≥6 months.
5. HER2-positive recurrent or metastatic BC patients who have received at most one anti-HER2 therapy after diagnosis;.
6. PD-L1-positive (cut-off ≥ 1% stained cells);
7. Patients with assessable target lesion as per RECIST 1.1 and irRECIST criteria.
8. ECOG PS score 0 or 1, estimated survival time ≥3 months, and can be followed-up.
9. Cardiopulmonary function is basically normal.
10. Liver function is basically normal.
11. Have sufficient baseline hematology parameters.
12. Coagulation Indicators: International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 times the upper limit of normal, unless drugs known to change INR and aPTT are used.
13. No history of serious heart, kidney and other important organs and endocrine disease.
14. Female patients of childbearing age have a negative pregnancy test and voluntarily take effective and reliable contraceptive measures.
15. The patients voluntarily signed an informed consent form.

Exclusion Criteria:

1. Participated in other clinical trials within 4 weeks;
2. Evidence of symptomatic central nervous system metastasis or pia mater disease.
3. History of receiving CD137 agonists or checkpoint blockade therapy (including anti-CD40, anti-CTLA-4, anti-PD-1, anti-PD-L1 monoclonal antibody therapy).
4. History of receiving paclitaxel for injection (Albumin Bound) in first-line chemotherapy for advanced disease.
5. History of autoimmune disease Including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease (IBD), etc.
6. Immunosuppressive drugs required within 2 weeks before enrollment or during this study. The following conditions are excluded: 1) intranasal, inhalation, topical or local steroid injection (e.g., intra articular injection); 2) physiological doses of systemic corticosteroids (≤ 10 mg/day prednisone or equivalent dose); 3) short term (≤ 7 days) use of steroids to prevent or treat non-autoimmune allergic diseases.
7. History of acute or chronic hepatitis B virus (HBV), or hepatitis C virus (HCV).
8. History of primary or acquired immunodeficiency (including HIV-positive).
9. History of hypersensitivity to the study medication
10. Pregnancy or lactation.
11. History of myocardial infarction within 6 months before enrollment, congestive heart failure (New York Heart Association [NYHA] Classes ≥ II), severe arrhythmia beyond drug control, or a decrease in LVEF to < 50% with previous trastuzumab neoadjuvant or adjuvant treatment.
12. History of other malignant disease within 5 years (except cured of in-situ carcinoma of the cervix, basal cell carcinoma of the skin and squamous cell carcinoma).
13. Participants who were judged by the investigator to be unsuitable for this study .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-12 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Assessed up to approximately 24 months
  PFS is defined as the time from the date of the first dose until first evidence of disease progression or death based on investigator assessment using RECIST 1.1 and irRECIST.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Assessed up to approximately 24 months
  ORR is defined as the percentage of participants who have a complete response (CR) or partial response (PR) based on CT/MRI, investigator assessment using RECIST 1.1 and irRECIST.
Clinical benefit rate (CBR) | Assessed up to approximately 24 months
  CBR is defined as the percentage of evaluable participants with best objective response of confirmed complete response or partial response per RECIST 1.1 and irRECIST, or prolonged stable disease (≥ 6 months).
Safety assessment (AEs and SAEs) | From the time of inform consent form signature until 30 days after end of treatment
  Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Director of Breast Cancer Section
Locations (1):
- Cancer Hospital Chinese Academy Of Medical Sciences, Beijing, China